CLINICAL TRIAL: NCT04665427
Title: Factors That Influence the Occurrence of Bile Leaks After Biliary Anastomosis Surgery
Brief Title: Factors Influencing Occurrence of Bile Leaks in Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oran 1 (Other)
Responsible Party: Principal Investigator, Anisse Tidjane, Associate Professor, University of Oran 1
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: UOran1_surgery_Bile_leak
Record Dates: First submitted 2020-11-29; First posted 2020-12-11 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Bile Leak; Anastomotic Leak Biliary; Biliary Tract Fistula
Keywords: hepatobiliary surgery; Morbidity; leak; anastomosis
MeSH Terms: conditions — Biliary Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient in whom a bilioenteric anastomosis is performed for any etiology. (Other): Patient in whom a bilioenteric anastomosis is performed for any etiology..
  Interventions: Other: bilioenteric anastomosis i

INTERVENTIONS:
Other: bilioenteric anastomosis i — The creation of communication between a bile duct and a segment of the digestive tract, often to restore a flow of bile in the digestive tract,
  Other Names: hepatico duodenostomy; hepaticojejunostomy

SUMMARY:
The objective of our study is to identify the factors influencing the occurrence of a biliary leak after performing surgery leading to the creation of a biliary anastomosis to any segment of the digestive tract.

DETAILED DESCRIPTION:
The objective of our study is to identify the factors influencing the occurrence postoperative of biliary leaks, Sex, Age, BMI, Bilirubin level, Protein level, and surgical technique (And other factors)are analyzed to study their influence on occurrence of postoperative biliary leak.

ELIGIBILITY:
Inclusion Criteria:

* Any patient who has undergone a surgical bilioenteric anastomosis for any etiology.

Exclusion Criteria:

* Any patient who has undergone a nonsurgical (endoscopic / radiological) bilioenteric anastomosis.
* Subjects under the age of 18. Years.
* Subjects who refused to participate in this study.
* Cases of biliary and pancreatic anastomoses performed during the same surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2020-11-18 (Actual); Primary Completion 2022-07-18 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
The occurrence of a bile leak in the postoperative period (Day 0 to Day 90). | From (day 0) of surgery to (day 90)
  Occurrence of a bile leak visible through a drain, through the wound, visible on the control radiology, or after the occurrence of a peritoneal collection or biliary peritonitis.

SECONDARY OUTCOMES:
Postoperative hospital stay | From (day 0) of surgery to (day 90)
  length of postoperative hospital stay
Mortality | From day 0 to day 90
  Mortality after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Benali Tabeti, Pr, Study Chair — University Oran1
Locations (1):
- Departmenet of hepatobiliary surgery, EHU-1st November 1954, Oran., Oran, Algeria

IPD SHARING:
Plan to Share IPD: No